CLINICAL TRIAL: NCT03706599
Title: Fever Infants and Therapeutic Education in Emergency Department
Acronym: D-FI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K170306J / AOR12065
Record Dates: First submitted 2018-09-28; First posted 2018-10-16 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fever therapeutic education session (Experimental): Therapeutic education session on fever
  Interventions: Behavioral: Therapeutic education on fever
- Control therapeutic education session (Placebo Comparator): Control therapeutic education session (on household accidents)
  Interventions: Behavioral: Therapeutic education on household accidents

INTERVENTIONS:
Behavioral: Therapeutic education on fever — Session for therapeutique education on fever
  Arms: Fever therapeutic education session
Behavioral: Therapeutic education on household accidents — Session for therapeutic education on household accidents
  Arms: Control therapeutic education session

SUMMARY:
To evaluate the effect of a therapeutic education session on fever versus a control education session on household accidents on the behavior and knowledge of families concerning the management of infant fever between day 4 and day 7 after the intervention

DETAILED DESCRIPTION:
Increased attendance at pediatric emergencies is observed in many countries. Fever, a frequent reason for consultation in pediatric emergencies, contributes to this phenomenon and is known to cause panic reactions in parents that are not justified by the actual state of the child. The accurate identification of families' lack of knowledge of fever has allowed us to develop a therapeutic education session, after which families should be able to properly care for a febrile child without excessive use of emergency services.

The hypothesis is that a therapeutic education session on fever in infancy, intended for parents, carried out in pediatric emergencies, after a consultation for febrile illness will allow:

* improve family behaviors and knowledge regarding fever in children.
* limit the number of new consultations to pediatric emergencies in the next 6 months.

The project takes place in two successive phases.

1. First phase, which is now completed, consisted of 4 stages:

   A. Semi-structured interviews conducted by an anthropologist with parents of children aged 3 months to 2 years who consulted pediatric emergencies for the reason "fever". The anthropologist questioned the families about their perceptions of the fever, the perceived origin, the fears associated with this symptom, the behavior adopted, the reasons for the consultation in these services:

   B. Development of a therapeutic education session for fever. This session was conceived from the data of the literature but also from the results of the semi-directive interviews, in particular to better correspond to the sociocultural characteristics of the families consulting in pediatric emergencies.

   C. Elaboration of a questionnaire to evaluate behaviors and knowledge, called "D-FI" questionnaire: the thematic cross-sectional analysis of the interviews led to the construction of a knowledge assessment questionnaire on the management of fever in infants by families. This questionnaire will assess the effectiveness of the therapeutic education intervention.

   D. Validation of the D-Fi questionnaire in a test population: the questionnaire was administered to "uneducated" parents in the management of fever and to health professionals. The results between these two groups were compared. Different aspects have been studied:
   * Reliability of the questionnaire.
   * Quality of each selected item
   * Internal validity
   * Calculation of a score to assess skills and knowledge on fever
2. The study reported at Clinical trial corresponds to the second phase of this project.

A randomized controlled trial will evaluate the impact of the therapeutic education session developed in Phase 1 on family behaviors and knowledge on fever compared to a control intervention. The intervention control will be a health education session on the prevention of domestic accidents. The D-Fi survey designed during the first phase will be used during this test. The recruitment of consulting patients in two different hospitals, namely the hospitals of Robert-Debré (Paris 19th) and Necker-Enfants Malades (Paris 15th), will widen the socio-cultural diversity of the population included in this project and improve the external validity of the study.

ELIGIBILITY:
Inclusion Criteria:

* Francophone family who consults for a febrile illness of their child (defined by a t °> 38 °) aged from 3 months to 2 years at the time of passage to pediatric emergencies Presence of at least one parent or guardian of the child

Exclusion Criteria:

* Presence of chronic pathology Family already included in the study

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Behavior and knowledge score of families obtain through answering D-FI (Decrease Fever Infants) survey | Day 4
  score D-FI survey :D-FI survey is a scale measuring behavior and knowledge of families on fever. Range from 0 (low score) to 10 (high score=better knowledge and behavior).

SECONDARY OUTCOMES:
Behavior and knowledge of families obtain through answering D-FI (Decrease Fever Infants) survey | 6 months
  score D-FI survey :D-FI survey is a scale measuring behavior and knowledge of families on fever. Range from 0 (low score) to 10 (high score=better knowledge and behavior).
Number of medical consultation unplanned | 6 months
Number of pediatric emergency consultation | 6 months
Number of suboptimal care and severe bacterial infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: François Angoulvant, MD, PhD, Principal Investigator — APHP
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No